CLINICAL TRIAL: NCT04384796
Title: Turkish Validity and Reliability Study of Infant Movement Motivation Questionnaire
Brief Title: Turkish Version of Infant Movement Motivation Questionnaire
Status: Completed | Type: Observational
Sponsor: Yeditepe University (Other)
Responsible Party: Sponsor
Other Study IDs: KAEK:899
Record Dates: First submitted 2020-05-08; First posted 2020-05-12 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Infant Development; Temperament; Early Intervention; Infant Behavior
MeSH Terms: conditions — Infant Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Purpose: It is the examination of the Infant Movement Motivation Questionnaire of the validity and reliability of Turkish.

Pretest: Participants were informed about the aims of the study and fill in a consent form. They filled in a paper version of the Turkish translation of the Infant Movement Motivation Questionnaire. The parents had to answer questions about the content and meaning of the IMMQ items and sociodemographic.

Validation Study: Participants were informed about the aims of the study and filled in a consent form. The questionnaires of the survey filled in at the early intervention center. About 30 minutes were needed to answer the 27 questions of the IMMQ, Ages and Stages Questionnaire, and sociodemographic.

DETAILED DESCRIPTION:
The period when human life activity most intense is the first years of life. Different practices such as voicing, speaking, sitting, walking, mental skills, communication, socializing acquire new skills. Infant Movement Motivation Questionnaire(IMMQ) 27-item scale that questions babies' discovery, activity, motivation, and adaptation skills in daily life activities through the parent. The scale was developed in 2012 by Samantha Doralp. As the scale provides information about how babies spend their time in their natural environment and the personal characteristics of babies, it was decided to carry out a validity and reliability study in the Turkish language, considering the early use of support programs in clinical use. The development of this scale shows the first step in understanding the role of baby characteristics in the movement development of babies in the first year of life. A good understanding of the link between baby characteristics and motor development can have a significant impact on planning interventions and can have a significant impact in ensuring that a particular environment is optimally tailored to the child's use and needs.

ELIGIBILITY:
• Volunteers who have babies with typical development between 0-12 months

Exclusion Criteria:

* Parents of babies with a neurological diagnosis
* Parents of babies with vision, hearing loss
* Parents of babies with a genetic and metabolic diagnosis

Max Age: 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Babies between 0-12 months who meet the working criteria.
Sampling Method: Non-Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-05-15 (Actual)

PRIMARY OUTCOMES:
Infant Movement Motivation Questionnaire | 12 months
  The survey assesses the willingness of the movement of babies between 0 and 12 months. The questionnaire includes 27 questions in 4 areas: "activity, exploratory behavior, motivation, adaptation". The questionnaire is answered on a five-point Likert scale by caregivers.

SECONDARY OUTCOMES:
Ages and Stages Questionnaire-2, (ASQ 2) | 12 months
  It is used to evaluate the development of babies from 3 months 0 days to 60 months with 19 different questionnaires customized by age. It evaluates five different areas: communication, gross motor, fine motor, problem-solving, personal-social.
  Each question is answered by the parent as Yes, Sometimes and No. In the calculation of the points, Yes is recorded as 10 points, Sometimes 5 points, and No, 0 points.

CONTACTS AND LOCATIONS:
Locations (1):
- Ebru Altunalan, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Doralp S, Bartlett D. Infant Movement Motivation Questionnaire: development of a measure evaluating infant characteristics relating to motor development in the first year of life. Infant Behav Dev. 2014 Aug;37(3):326-33. doi: 10.1016/j.infbeh.2014.04.002. Epub 2014 May 28. PMID 24861943
- [Background] Doralp S, Bartlett DJ. Environmental opportunities questionnaire: development of a measure of the environment supporting early motor development in the first year of life. Disabil Rehabil. 2013 Sep;35(20):1692-7. doi: 10.3109/09638288.2012.751133. Epub 2013 Jan 25. PMID 23350756
- [Background] Cacola PM, Gabbard C, Montebelo MI, Santos DC. Further Development and Validation of the Affordances in the Home Environment for Motor Development-Infant Scale (AHEMD-IS). Phys Ther. 2015 Jun;95(6):901-23. doi: 10.2522/ptj.20140011. Epub 2014 Dec 18. PMID 25524875